CLINICAL TRIAL: NCT05534685
Title: To Compare the Effect of Intratracheal Administration of Surfactant vs. Surfactant/Budesonide on the Incidence of Bronchopulmonary Dysplasia in Preterm Infants Less Than 34 Weeks of Gestation
Brief Title: Budesonia + Intratracheal Surfactant in Incidence of Bronchopulmonary Dysplasia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Collaborators: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, Guadalupe Gómez Rodríguez, principal investigator, Instituto Mexicano del Seguro Social
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Budesonia + surfactan
Record Dates: First submitted 2022-09-06; First posted 2022-09-09 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Respiratory Tract Diseases
Keywords: Surfactant/Budesonide, Bronchopulmonary Dysplasia. Preterm
MeSH Terms: conditions — Respiratory Tract Diseases | interventions — Budesonide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intratracheal administration of surfactant/budesonide on the incidence of bronchopulmonary dysplasia (Experimental): Group A will be given surfactant (beractant, lung phospholipids of bovine origin. Injectable suspension 1ml contains 25mg) at a dose of 100mg/kg or 4ml/kg and budesonide (budesonide, nebulized suspension 2ml contains 0.500mg) at a dose of 0.250 mg/kg or 1 ml/kg.
  Interventions: Other: intratracheal administration of surfactant/budesonide
- intratracheal administration of surfactant on the incidence of bronchopulmonary dysplasia (Experimental): Group B will receive surfactant alone (beractant, lung phospholipids of bovine origin. Injectable suspension 1ml contains 25mg) administered at a dose of 100mg/kg or 4ml/kg.
  Interventions: Other: incidence of bronchopulmonary dysplasia

INTERVENTIONS:
Other: intratracheal administration of surfactant/budesonide — 328 patients will be included from Group A: 164 patients, from Group B: 164 patients who meet the selection criteria within the first 4 hours of hospital stay, after the authorization of the parents or guardian signing the informed consent. According to the assigned group, the preparation of surfactant or surfactant/budesonide in the syringe will be carried out, prior to performing the tracheal cannulation procedure. Group A will be given surfactant (beractant, lung phospholipids of bovine origin. Injectable suspension 1ml contains 25mg) at a dose of 100mg/kg or 4ml/kg and budesonide (budesonide, nebulized suspension 2ml contains 0.500mg) at a dose of 0.250 mg/kg or 1 ml/kg. Group B will receive surfactant alone (beractant, lung phospholipids of bovine origin. Injectable suspension 1ml contains 25mg) administered at a dose of 100mg/kg or 4ml/kg.
  Other Names: intratracheal administration of surfactant
  Arms: intratracheal administration of surfactant/budesonide on the incidence of bronchopulmonary dysplasia
Other: incidence of bronchopulmonary dysplasia — . Subsequently, follow-up will be carried out at 12 hours to assess the administration of the second dose of surfactant, type of mechanical ventilation, inspired fraction of oxygen (Fi02), arterial pressure of oxygen (PaO2), partial pressure of carbon dioxide (PaCO2 ), mean airway pressure (PMVA), oxygen index (IO), oxygen saturation by pulse oximetry, weekly follow-up of the patient will continue for 28 days, evaluating the same parameters to make a diagnosis of bronchopulmonary dysplasia and finally at 36 postmenstrual weeks of gestation in those under 32 SDG or at discharge and at 56 postmenstrual days of life in those over 32 SDG or at discharge, allowing the severity of the disease to be determined
  Arms: intratracheal administration of surfactant on the incidence of bronchopulmonary dysplasia

SUMMARY:
Objectiv: To compare the effect of intratracheal administration of surfactant vs. surfactant/budesonide on the incidence of bronchopulmonary dysplasia in preterm infants less than 34 weeks of gestation.

Material and methods: Study design: Double-blind randomized controlled clinical trial.Inclusion criteria: Newborns under 34 weeks of gestation with a diagnosis of Respiratory Distress Syndrome requiring administration of surfactant, invasive and/or non-invasive ventilatory support admitted to the Neonatal Intensive Care Unit service and pathological nursery. Procedure: 328 patients will be included from Group A: 164 patients, from Group B: 164 patients who meet the selection criteria within the first 4 hours of hospital stay, after the authorization of the parents or guardian signing the informed consent. According to the assigned group, the preparation of surfactant or surfactant/budesonide in the syringe will be carried out, prior to performing the tracheal cannulation procedure. Group A will be given surfactant (beractant, lung phospholipids of bovine origin. Injectable suspension 1ml contains 25mg) at a dose of 100mg/kg or 4ml/kg and budesonide (budesonide, nebulized suspension 2ml contains 0.500mg) at a dose of 0.250 mg/kg or 1 ml/kg. Group B will receive surfactant alone (beractant, lung phospholipids of bovine origin. Injectable suspension 1ml contains 25mg) administered at a dose of 100mg/kg or 4ml/kg. Subsequently, follow-up will be carried out at 12 hours to assess the administration of the second dose of surfactant, type of mechanical ventilation, inspired fraction of oxygen (Fi02), arterial pressure of oxygen (PaO2), partial pressure of carbon dioxide (PaCO2 ), mean airway pressure (PMVA), oxygen index (IO), oxygen saturation by pulse oximetry, weekly follow-up of the patient will continue for 28 days, evaluating the same parameters to make a diagnosis of bronchopulmonary dysplasia and finally at 36 postmenstrual weeks of gestation in those under 32 SDG or at discharge and at 56 postmenstrual days of life in those over 32 SDG or at discharge, allowing the severity of the disease to be determined.Sample size: The study includes an intervention group (surfactant/budesonide group) and a control group (surfactant only group), each with 164 patients, for a total of 328 patients.

Statistical analysis: The Chi-Square statistician will be used with a precision requirement of 95%, where p<=0.05. The risk measurement will be with RR (RR) and its 95% confidence interval (CI). NICSS 2007 statistical package will be used.

Ethical aspects: This study must have an authorization signature through informed consent.

DETAILED DESCRIPTION:
MATERIAL AND METHODS STUDY DESIGN Clinical, controlled, randomized, double-blind trial.

PLACE WHERE THE STUDY WILL BE DEVELOPED The study will be carried out in the High Specialty Medical Unit No. 48 of the Mexican Institute of Social Security of the CMN of Bajío León Guanajuato, in the Neonatal Intensive Care Unit (NICU) and pathological nursery service.

Location: Av. Mexico and Insurgentes S/N Col. Los Paraisos, CP 37220

DURATION OF THE STUDY Once authorized by the CNIC, the study will be carried out until the indicated sample is completed.

SOURCE OF INFORMATION Clinical records of all patients who enter the study in the NICU and pathological nursery service

PARTICIPANTS:

Preterm newborn patients under 34 SDG, both sexes, beneficiaries of the Mexican Institute of Social Security UMAE 48, who have a clinical and radiological diagnosis of respiratory distress syndrome and require the administration of surfactant as treatment.

TYPE OF SAMPLING Simple random without replacement

SAMPLE SIZE: It was determined in relation to a study carried out in Taiwan by Tsu F. et al. in the year 2016. The formula is used to compare two groups with different proportions (50% vs 29%) with a sample of the same size to obtain a two-tailed alpha of .05 and a minimum power of 80%, an OR is necessary of 0.409 or RR of .58 and Z alpha values of 1.96 and Z beta of .8416 with a combined proportion of .395.

A = Zα√P(1-P)(1/q1 + 1/q0) = 1.9163

B = Zβ√P1(1-P1)(1/q1) + P0(1-P0)(1/q0) = 0.8036

C = (P1-P0)2 = 0.0441

Total group size = N = (A+B)2/C = 168

The study includes an intervention group (surfactant/budesonide group) and a control group (surfactant group), each of them with 168 patients, with a total of 336 patients, 20% is added for the expected losses of patients.

SELECTION CRITERIA

• Inclusion criteria: Newborns less than 34 weeks of gestation and weighing less than 1500-2000g. Newborns less than 32 weeks of gestation and weighing less than 750-1500g Preterm newborn with clinical and radiographic data of respiratory distress syndrome requiring administration of surfactant.

Newborn both sexes. Preterm newborn requiring invasive and/or non-invasive ventilatory support. Preterm infant who has and does not have antenatal exposure to steroids. • Exclusion criteria: Patient with major congenital malformations, term newborn

• Elimination criteria: Patient whose parents withdraw their consent.

VARIABLES

Independent variable:

Administration of surfactant/budesonide

Dependent variable:

bronchopulmonary dysplasia

Covariates:

ENSURE VS MITS Technique

STATISTIC ANALYSIS Student's t test or Mann Whitney U test will be performed for differences in means regarding the general characteristics of the patients, for continuous variables, the mean values of each moment of each group for variables such as FiO2, PO2, PCO2, pH, oxygenation index and Mean airway pressure were derived from a generalized linear model with generalized estimation equations and difference values over time, the Chi-Square or Fisher exact statistician for categorical variables such as mortality and morbidity with a precision requirement of 95%, where p<=0.05. The risk measurement will be with relative risk (RR) and its confidence interval (CI) of 95%. NICSS 2007 statistical package will be used.

PROCEDURES After approval by the National Committee for Scientific Research (CNIC).

The researchers responsible for the patient registry are:

Dr. Guadalupe Gómez Rodríguez, Dr. Evaldo Jesús Rodríguez Mejía. On a daily basis, the patients who meet the selection criteria will be identified within the first 2 to 4 hours of the patient's hospital stay, the parents or guardians will be contacted personally and they will be invited to participate in the study, explaining them fully and in detail. possible that it is bronchopulmonary dysplasia and why it occurs, what the study consists of, its objectives, its risks and benefits, and if they agree to participate, they will be asked to sign the informed consent letter; If they do not agree to participate, it will be made clear to them that this will not affect the type of care they receive in the hospital unit. Informed consent will be obtained by collaborating physicians at different times: Dr. Fátima de Rosario Estrada Pacheco (morning shift), Dr. Edgar Ulises Sanvicente Santoscoy (evening shift), Dr. Fátima de Rosario Estrada Pacheco (morning shift) , Dr. Eduardo Isaac Rodríguez Rodríguez (Monday, Wednesday and Friday night shift), Marco Antonio Guerrero Zúñiga (Tuesday, Thursday and Sunday night shift). It will be performed during the first 2 to 4 hours of the patient's life (considering this time pertinent for the administration of treatment for respiratory distress syndrome).

Randomization and blinding:

The hidden randomization will be generated by means of cards elaborated based on the random tables see annex (2), the cards will be elaborated and placed in closed envelopes available only for the head of the service, treating physician, resident who will deliver them to the corresponding nurse, in such a way that the doctor and the patient will not know if they belong to the experimental group or the control group. The nursing service will be responsible for preparing and providing the physician with the surfactant plus budesonide (group A), which is the experimental group, or the surfactant alone (group B), which is the control group.

The patient must have a clinical and radiographic diagnosis of RDS and the need for administration of surfactant issued by the treating physician and collaborator of the study will be assessed in accordance with the European RDS Guide 2019. (6) Once the patient is assigned to a study group, the intervention will be carried out, which consists of the administration of surfactant plus budesonide (Group A) or surfactant alone (Group B), according to the randomization system.

The administration of the medication(s) will be carried out by the collaborating neonatologists and those responsible for the patient:

Dr. Edgar Ulises Sanvicente Santoscoy, Dr. Fátima de Rosario Estrada Pacheco, Dr. Eduardo Isaac Rodríguez Rodríguez, Dr. Marco Antonio Guerrero Zúñiga assigned neonatologists from the NICU, pathological nursery and obstetrics surgery area, which belong to UMAE No. 48 of the IMSS .

Surfactant (Beractant, lung phospholipids of bovine origin. Injectable suspension 1ml contains 25 mg) will be administered in group A at a dose of 100 mg/kg or 4 ml/kg and budesonide (budesonide, nebulized suspension 2ml contains 0.500 mg) at a dose of 0.250 mg/kg or 1 ml/kg. If you belong to group B, you will receive surfactant alone (beractant, lung phospholipids of bovine origin. Injectable suspension 1ml contains 25mg) administered at a dose of 100mg/kg or 4ml/kg every 12h.

For the administration of the medications, prior asepsis and antisepsis will be carried out, placement of sterile fields, direct laryngoscopy, cannulation of the trachea to subsequently carry out the instillation (drop by drop a liquid in a specific site) of the or medications. The procedure may be performed using the INSURE technique, which consists of intubating the patient, administering the surfactant or surfactant/budesonide and extubating immediately, or by the MIST technique, which consists of administering the surfactant or surfactant/budesonide through a endotracheal semi-rigid vascular catheter

ELIGIBILITY:
Inclusion Criteria:

* Preterm newborn with clinical and radiographic data of respiratory distress syndrome requiring administration of surfactant.

Newborn both sexes. Preterm newborn requiring invasive and/or non-invasive ventilatory support. Preterm infant who has and does not have antenatal exposure to steroids.

Exclusion Criteria:Patient with major congenital malformations, term newborn

• Elimination criteria: Patient whose parents withdraw their consent.

Ages: 26 Weeks to 34 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 336 (Estimated)
Dates: Start 2022-09-20 (Estimated); Primary Completion 2023-02-20 (Estimated); Study Completion 2023-07-20 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Treatment-Related Adverse Events | the fisrt 48 hours, util the week of extrauterine will be monitored
  evaluate the adverse events that occur. Budesonide: headache, stomach pain, hyperglycemia, electrolyte disturbances. Surfactant: bradycardia, hypotension, endotracheal tube obstruction, desaturation, patent ductus arteriosus, pulmonary hemorrhage

SECONDARY OUTCOMES:
Assess the indicence of broncopulmonary displasia | first 28 days of extrauterine life our 36 postmenstrual weeks of gestation
  At 12 hours, it will be recorded if the patient required a second dose of surfactant and the date and time, type of mechanical ventilation, inspired fraction of oxygen (Fi02), arterial blood gases will be taken to analyze arterial oxygen pressure (PaO2), pressure partial carbon dioxide (PaCO2), mean airway pressure (PMVA), oxygen index (IO), oxygen saturation by pulse oximetry. Weekly follow-up of the patient will continue for 28 days, evaluating the same parameters to make a diagnosis of bronchopulmonary dysplasia and finally at 36 postmenstrual weeks of gestation in those under 32 SDG or at discharge and at 56 postmenstrual days of life in those over 32 SDG or at discharge, allowing to determine the severity of the disease.

CONTACTS AND LOCATIONS:
Overall Officials: Guadalupe Gómez Rodríguez, Principal Investigator — Instituto Mexicano del Seguro Social; José Luis Felipe Luna Anguiano, Study Director — Instituto Mexicano del Seguro Social

REFERENCES:
- [Result] Tang W, Chen S, Shi D, Ai T, Zhang L, Huang Y, Fan Y, Du Y. Effectiveness and safety of early combined utilization of budesonide and surfactant by airway for bronchopulmonary dysplasia prevention in premature infants with RDS: A meta-analysis. Pediatr Pulmonol. 2022 Feb;57(2):455-469. doi: 10.1002/ppul.25759. Epub 2021 Nov 25. PMID 34783192
- [Result] Gharehbaghi MM, Mhallei M, Ganji S, Yasrebinia S. The efficacy of intratracheal administration of surfactant and budesonide combination in the prevention of bronchopulmonary dysplasia. J Res Med Sci. 2021 May 27;26:31. doi: 10.4103/jrms.JRMS_106_19. eCollection 2021. PMID 34345242